CLINICAL TRIAL: NCT06178978
Title: Device for Monitoring Age-related Macular Degeneration (AMD)
Brief Title: Device for Age-related Macular Degeneration (AMD)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yannis Paulus, Associate Professor, Department of Ophthalmology and Visual Sciences, University of Michigan
Other Study IDs: HUM00187177
Record Dates: First submitted 2023-08-24; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Age-Related Macular Degeneration
Keywords: age-related macular degeneration; macular degeneration; AMD; Home monitoring
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age-related macular degeneration: Patients with age-related macular degeneration.
  Interventions: Device: KalEYEdoscope

INTERVENTIONS:
Device: KalEYEdoscope — KalEYEdoscope is a digital, handheld device utilizing shape-discrimination hyperacuity to distinguish the severity of age-related macular degeneration. In the future, developing such a device for home monitoring of macular degeneration may increase access to timely treatment to prevent vision loss.
  This study was conducted at the Kellogg Eye Center in Ann Arbor. Participants in the outpatient setting who agreed to enroll in the study tested the device and provided user feedback via a questionnaire as well as completed questionnaires about their visual function. This study assessed the usability, comfort, duration, ergonomics, and ease of use of the device among AMD patients in a single session.

SUMMARY:
This study involves user acceptability and feedback of KalEYEdoscope, a digital, handheld device utilizing shape-discrimination hyperacuity to distinguish the severity of age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This is a patient-experience study being conducted at the Kellogg Eye Center in Ann Arbor in the outpatient setting. Patients who agree to enroll in the study will test the device and provide user feedback via a questionnaire as well as complete questionnaires about their visual function. The preliminary study looks at the usability of using this device for monitoring of age-related macular degeneration, obtaining user feedback to enhance the design. In the future, developing such a device for home monitoring of macular degeneration may increase access to timely treatment to prevent vision loss.

To gather user feedback on a digital, non-invasive, handheld device in the outpatient AMD patient population, with the goal of developing a user-friendly, portable device to monitor AMD progression, this study assesses the usability, comfort, duration, ergonomics, and ease of use of the device among AMD patients in a single session.

Data collected during the test may include but is not limited to the length of the test, boot time, screen transition time. The participants will then fill out the Visual Function Questionnaire-25, the System Usability Scale (SUS), and may include targeted questions designed by the study team to evaluate the participant experience with the device and visual function.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18 years or older with age-related macular degeneration who is seen at the Kellogg Eye Center.

Exclusion Criteria:

* pregnant women, prisoners, severe cognitive impairment, and diagnoses (mental or neuromuscular disorders) which could preclude independent use of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
System usability scale | immediate during a single office visit - generally 5- 15 minutes
  Obtain user feedback via a questionnaire and evaluate the usability of using this device.

SECONDARY OUTCOMES:
National Eye Institute Visual function questionnaire (NEI VFQ 25) | immediate during a single office visit - generally 5- 15 minutes
  Participants complete 25-question questionnaire about their visual function.
Participant Experience Survey | immediate during a single office visit - generally 5- 15 minutes
  Participants complete 8 qualitative questions with a Likert scale about the device and using the device.

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Paulus, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
HIPAA compliant data sharing